CLINICAL TRIAL: NCT02248779
Title: Assessing Insulin Sensitivity and Diabetes Risk in Childhood Cancer Survivors Treated With Abdominal Irradiation: A Pilot Study
Brief Title: Assessing Insulin Sensitivity and Diabetes Risk in Childhood Cancer Survivors Treated With Abdominal Irradiation
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-202
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Childhood Cancer Survivors Treated With Abdominal Radiation
Keywords: Diabetes Risk; 14-202

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood

GROUPS / COHORTS (2):
- treated < 20 years prior to study enrollment: The following information will be gathered:
  A. Height, weight, waist circumference, blood pressure B. Oral glucose tolerance testing (OGTT) where in participants will ingest a standard oral glucose load (75 grams) in liquid formulation after an overnight fast. Blood samples for glucose and insulin concentrations will be taken at 0, 30, 60, 90, and 120 minutes post-glucose load.
  C. Glutamic acid decarboxylase (GAD), islet cell (ICA-512), and insulin autoantibody (IAA) titers as well as serum adiponectin and hemoglobin A1c.
  All enrolled patients will have a discussion with an LTFU doctor regarding the results of testing. Counseling and referral to a specialist will be provided if indicated.
- treated ≥ 20 years prior to study enrollment: The following information will be gathered:
  A. Height, weight, waist circumference, blood pressure B. Oral glucose tolerance testing (OGTT) where in participants will ingest a standard oral glucose load (75 grams) in liquid formulation after an overnight fast. Blood samples for glucose and insulin concentrations will be taken at 0, 30, 60, 90, and 120 minutes post-glucose load.
  C. Glutamic acid decarboxylase (GAD), islet cell (ICA-512), and insulin autoantibody (IAA) titers as well as serum adiponectin and hemoglobin A1c.
  All enrolled patients will have a discussion with an LTFU doctor regarding the results of testing. Counseling and referral to a specialist will be provided if indicated.

SUMMARY:
The purpose of this study is to better understand the risk factors and causes of diabetes in people who received radiation to the abdomen as children. The investigators hope this information will allow them to improve how they screen people at risk for diabetes and how they treat patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of childhood cancer between 0-21 years of age
* Prior treatment with abdominal radiation at MSKCC
* Two or more years from completion of therapy
* Records of cancer diagnosis and treatment (including radiation records) available

Exclusion Criteria:

* Known diagnosis of diabetes
* Previous treatment with any radiation impacting the brain (cranial radiation, craniospinal radiation, total body irradiation)
* Neurocognitive deficits that impair ability to give informed consent or assent
* Patients predicted to have difficult intravenous access, who will likely require multiple venipuncture attempts

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Childhood cancer survivors followed by the Pediatric Long-Term Follow-Up Program or Adult Long-Term Follow-Up Program will be recruited for the current study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-09-22 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
characterize β cell function | 2 years
  we will be able to estimate the proportion of patients with abnormalities of insulin sensitivity or β cell function, as assessed by the OGTT, to within ± 0.14.
insulin sensitivity | 2 years
  we will be able to estimate the proportion of patients with abnormalities of insulin sensitivity or β cell function, as assessed by the OGTT, to within ± 0.14.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle N. Friedman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/